CLINICAL TRIAL: NCT03323112
Title: Immune Responses to Influenza Vaccinations and Viruses Among Health Care Personnel
Brief Title: Immune Responses in Health Care Personnel
Status: Recruiting | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Sponsor
Other Study IDs: FinFLU_HCPimmu_2017THL
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Influenza
Keywords: influenza; vaccination; health care workers; immune responses; humoral immunity; cellular immunity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples, PBMC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza vaccine recipients: Health care workers vaccinated by their occupational health care according to the routine praxis.
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — Vaccine for prevention of influenza. Vaccines change by influenza season.

SUMMARY:
This is an investigator-initiated 10 year long open cohort observational study, aiming to increase the understanding of the humoral and cellular immunological mechanisms of vaccination against influenza, including effects of repeated vaccination, the duration of protection, immunity against circulating viruses, as well as factors affecting the immunological responses and immunity against other vaccine preventable infectious diseases among health care personnel.

DETAILED DESCRIPTION:
Influenza vaccination is given according to the normal routine of Hospital District of Helsinki and Uusimaa (HUS) occupational health care. Blood samples will be collected before vaccination, 5 weeks after vaccination and 6 months after vaccination. Both the same participants and also new participants will be recruited each year. The analysis will be mainly descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Members of health care or laboratory personnel in HUS having decided to take the seasonal influenza vaccination by the routine occupational health care service
* General good health as established by or volunteer's own statement
* Written informed consent
* Presumably able and willing to participate in the study during the starting influenza season

Exclusion Criteria:

* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Administration (longer than 14 days) of immunosuppressants or other immune- modifying drugs within 6 months before the vaccination; oral corticosteroids in dosages of 20 mg/day or more prednisolone or equivalent are excluded; inhaled or topical steroids are allowed.
* Pregnancy or lactation
* Acute disease at the time of enrolment (defined as the presence of a moderate or severe illness with or without fever)
* Contraindication for influenza vaccination
* Any other criteria which, in the investigator's or dedicated study staff member's opinion, would compromise the ability of a subject to participate in the study, a subject's well-being, or the outcome of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health care professionals affiliated by HUS
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2027-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Humoral immunity against each present season's vaccine and circulating influenza strains | 10 years
  The presence and titer of antibodies against circulating influenza virus strains and vaccine strains of the current season from pre- and post-vaccination serum samples

SECONDARY OUTCOMES:
Humoral immunity against previous seasons' vaccine and circulating influenza strains | 10 years
  To assess the presence and titer of antibodies to circulating influenza strains and vaccine virus strains of previous seasons from pre- and post-vaccination serum samples
Cellular immunity against current and previous seasons' vaccine and circulating influenza strains | 10 years
  The cellular immune responses to circulating influenza viruses and vaccine strains of the current and previous seasons from pre- and post-vaccination peripheral blood mononuclear cells (PBMCs) and cell culture supernatants
Effect of repeated vaccination against influenza | 10 years
  The effect of the number of previous influenza vaccinations on the quality and quantity of Humoral and cellular immunity to circulating influenza strains and vaccine strains of the current and previous seasons

OTHER OUTCOMES:
Factors affecting humoral and/or cellular immune responses to influenza viruses or vaccination | 10 years
  Exploration of biological or chemical factors that are/will be known or suspected to affect the humoral and/or cellular immune responses to influenza viruses or vaccination
Immunity against other microbes causing vaccine preventable diseases among health care workers | 10 years
  Assessment of humoral and cellular immunity to microbes other than influenza virus causing vaccine preventable diseases
Developing methods to measure immunity against vaccine preventable diseases | 10 years
  developing laboratory methodologies to assess immunity to influenza and other microbes causing vaccine preventable diseases

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Nohynek, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- The Hospital District of Helsinki and Uusimaa, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No